CLINICAL TRIAL: NCT00375388
Title: Study of Metformin HCL in Patients With Type 2 Diabetes Intensively Treated With Insulin: a Treatment Strategy for Insulin Resistance in Type 2 Diabetes Mellitus: a Randomized Controlled Trial
Brief Title: The HOME Trial: Hyperinsulinaemia: the Outcome of Its Metabolic Effects, a Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bethesda General Hospital, Hoogeveen (Other)
Collaborators: Takeda (Industry); LifeScan (Industry); Merck KGaA, Darmstadt, Germany (Industry); Dupont Merck (Industry); Merck Sharp & Dohme LLC (Industry); Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MET/NL/97.01
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Metformin on top of insulin therapy; Randomized placebo-controlled trial; Diabetes regulation; Daily dose of insulin; Body Weight; Patients with type 2 diabetes; Intensive insulin therapy; Age: 30-80 years; Body mass index; Lipids; Blood Pressure; Endothelial function; Low grade inflammation; Fibrinolysis; Microvascular complications; Macrovascular complications
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Body Weight

INTERVENTIONS:
Drug: Metformin on top of intensive insulin therapy

SUMMARY:
The HOME-trial is a prospective, randomized controlled trial. The purpose of this study is to investigate the effects of metformin HCL in patients with type 2 diabetes mellitus intensively treated with insulin on the quality of the metabolic control of diabetes, the daily dose of insulin, the lipid profile, the blood pressure, the incidence / progression of microvascular and macrovascular complications, and on the qualify of life (Diabetes Health Profile). Early results had been published in Diabetes Care, December 2002, pages 2133-2140.

DETAILED DESCRIPTION:
The HOME-trial is a prospective, randomized controlled trial. The purpose of this study is to investigate the effects of metformin HCL in patients with type 2 diabetes mellitus intensively treated with insulin on the quality of the metabolic control of diabetes, the daily dose of insulin, the lipid profile, the blood pressure, the incidence / progression of microvascular and macrovascular complications, and on the qualify of life (Diabetes Health Profile). Early results had been published in Diabetes Care, December 2002, pages 2133-2140.

Phase: Phase III

Study Type: Interventional

Overall Status: No longer recruiting (all patients have finished the study)

Study Start Date 02 January 1998

Study Completion Date October 2002

Study Design:

Study Purpose: Treatment Allocation: 1 randomized 0 non randomized Masking: Double blind Control: Placebo Assignment: Parallel Endpoints: Safety / Efficacy

Primary Outcome:

• To investigate the quality of the metabolic control of diabetes and related variables (daily dose of insulin, body weight).

Secondary Outcome:

* To investigate the occurrence of macro- and microvascular complications.
* To investigate the quality of life and to perform a socio-economic evaluation.

Conditions:

Type 2 diabetes mellitus requiring insulin therapy.

Keywords:

Type 2 diabetes mellitus; metformin; randomized; double-blind; placebo-controlled; diabetes regulation

Interventions: Metformin (850 mg) or placebo 1-3 times daily.

Insulin: 4 times daily or 'mixtures' of 30% rapidly and 70% slowly acting insulin, 2 times daily.

Eligibility Criteria (only add main ones)

Inclusion Criteria:

* Patients of both sexes (women after menopause, women of child-bearing age after sterilization or if practicing reliable contraception)
* Type 2 DM requiring insulin therapy after failure of maximal oral antidiabetic treatment (glycosylated Hb > 7.5%) and need for exogenous insulin. (No concomitant use of oral antidiabetic agents)
* Being ambulatory
* Age: 30 to 80 years
* Proven absence of Islet Antibodies, if QI < 28 kg/m2
* Insulin therapy 4 times daily (21), or insulin therapy 2 times daily using insulin 'mixtures' (rapidly and slowly acting)
* Standard dietary prescription by the dietician
* Absence of keto-acidosis
* Informed consent

Exclusion Criteria:

* Congestive heart failure, NYHA-classes III or IV
* Cardiac failure and/or myocardial infarction in the last four months before enrolment
* Other severe organic / systemic disease
* Metformin-induced lactic-acidosis
* Intolerance to metformin hydrochloride
* Renal disease or renal dysfunction
* Hypoxic states
* Severe hepatic dysfunction
* Excessive alcohol intake, acute or chronic
* Acute or chronic metabolic acidosis

Gender: Both

Age: 30 - 80 years

Target Number of Subjects: 400 (200 metformin, 200 placebo)

Central Contact:

Name: Adriaan Kooy , internist - diabetologist Degree: MD, PhD Phone: 0528-286222 Extension: 624 Mail: kooy.a@bethesda.nl

Study Official/ Investigators Name: Adriaan Kooy Degree: MD, PhD Officials Role: Study Principal Investigator

Organizational Affiliation:

Bethesda Hospital Hoogeveen Dr. G.H. Amshoffweg 1 7909 AA Hoogeveen The Netherlands

Locations:

Facility: Bethesda Hospital Hoogeveen City: Hoogeveen State/Province: Drenthe Country: The Netherlands Recruitment Status: No longer recruiting (all patients finished)

Facility: Diaconesses' Hospital Meppel City: Meppel State/Province: Drenthe Country: The Netherlands Recruitment Status: No longer recruiting (all patients finished)

Facility: Hospital Coevorden - Hardenberg City: Coevorden State/Province: Drenthe Country: The Netherlands Recruitment Status: No longer recruiting (all patients finished)

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes (women after menopause, women of child-bearing age after sterilization or if practicing reliable contraception)
* Type 2 DM requiring insulin therapy after failure of maximal oral antidiabetic treatment (glycosylated Hb > 7.5%) and need for exogenous insulin. (No concomitant use of oral antidiabetic agents)
* Being ambulatory
* Age: 30 to 80 years
* Proven absence of Islet Antibodies, if QI < 28 kg/m2
* Insulin therapy 4 times daily (21), or insulin therapy 2 times daily using insulin 'mixtures' (rapidly and slowly acting)
* Standard dietary prescription by the dietician
* Absence of keto-acidosis
* Informed consent

Exclusion Criteria:

* Congestive heart failure, NYHA-classes III or IV
* Cardiac failure and/or myocardial infarction in the last four months before enrolment
* Other severe organic / systemic disease
* Metformin-induced lactic-acidosis
* Intolerance to metformin hydrochloride
* Renal disease or renal dysfunction
* Hypoxic states
* Severe hepatic dysfunction
* Excessive alcohol intake, acute or chronic
* Acute or chronic metabolic acidosis

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 1998-01; Study Completion 2002-10

PRIMARY OUTCOMES:
To investigate the quality of the metabolic control of diabetes and related variables (daily dose of insulin, body weight).

SECONDARY OUTCOMES:
To investigate the occurrence and progression of macro- and microvascular complications.
To investigate the quality of life.
To perform a socio-economic evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Adriaan Kooy, MD, PhD, Principal Investigator — Bethesda General Hospital and Bethesda Diabetes Center, Hoogeveen, The Netherlands (for address: see above); Coen Stehouwer, MD, PhD, Study Director — University Hospital of Maastricht, The Netherlands
Locations (1):
- Bethesda General Hospital and Bethesda Diabetes Center, Hoogeveen, Drenthe, Netherlands

REFERENCES:
- [Result] Wulffele MG, Kooy A, Lehert P, Bets D, Ogterop JC, Borger van der Burg B, Donker AJ, Stehouwer CD. Combination of insulin and metformin in the treatment of type 2 diabetes. Diabetes Care. 2002 Dec;25(12):2133-40. doi: 10.2337/diacare.25.12.2133. PMID 12453950
- [Derived] Stultiens JMG, Top WMC, Kimenai DM, Lehert P, Bekers O, Stehouwer CDA, Kooy A, Meex SJR. Metformin and high-sensitivity cardiac troponin I and T trajectories in type 2 diabetes patients: a post-hoc analysis of a randomized controlled trial. Cardiovasc Diabetol. 2022 Apr 4;21(1):49. doi: 10.1186/s12933-022-01482-z. PMID 35379238
- [Derived] Out M, Becker ML, van Schaik RH, Lehert P, Stehouwer CD, Kooy A. A gene variant near ATM affects the response to metformin and metformin plasma levels: a post hoc analysis of an RCT. Pharmacogenomics. 2018 Jun 1;19(8):715-726. doi: 10.2217/pgs-2018-0010. Epub 2018 May 23. PMID 29790415
- [Derived] Out M, Top WMC, Lehert P, Schalkwijk CA, Stehouwer CDA, Kooy A. Long-term treatment with metformin in type 2 diabetes and vitamin D levels: A post-hoc analysis of a randomized placebo-controlled trial. Diabetes Obes Metab. 2018 Aug;20(8):1951-1956. doi: 10.1111/dom.13327. Epub 2018 May 14. PMID 29667290
- [Derived] Out M, Kooy A, Lehert P, Schalkwijk CA, Stehouwer CDA. Long-term treatment with metformin in type 2 diabetes and methylmalonic acid: Post hoc analysis of a randomized controlled 4.3year trial. J Diabetes Complications. 2018 Feb;32(2):171-178. doi: 10.1016/j.jdiacomp.2017.11.001. Epub 2017 Nov 8. PMID 29174300
- [Derived] Out M, Miedema I, Jager-Wittenaar H, van der Schans C, Krijnen W, Lehert P, Stehouwer C, Kooy A. Metformin-associated prevention of weight gain in insulin-treated type 2 diabetic patients cannot be explained by decreased energy intake: A post hoc analysis of a randomized placebo-controlled 4.3-year trial. Diabetes Obes Metab. 2018 Jan;20(1):219-223. doi: 10.1111/dom.13054. Epub 2017 Sep 14. PMID 28681986
- [Derived] de Jager J, Kooy A, Lehert P, Wulffele MG, van der Kolk J, Bets D, Verburg J, Donker AJ, Stehouwer CD. Long term treatment with metformin in patients with type 2 diabetes and risk of vitamin B-12 deficiency: randomised placebo controlled trial. BMJ. 2010 May 20;340:c2181. doi: 10.1136/bmj.c2181. PMID 20488910
- [Derived] Kooy A, de Jager J, Lehert P, Bets D, Wulffele MG, Donker AJ, Stehouwer CD. Long-term effects of metformin on metabolism and microvascular and macrovascular disease in patients with type 2 diabetes mellitus. Arch Intern Med. 2009 Mar 23;169(6):616-25. doi: 10.1001/archinternmed.2009.20. PMID 19307526